CLINICAL TRIAL: NCT03351621
Title: The Reality of Nutritional Therapy in Brazil: Quality Assessment
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Professor, Federal University of Minas Gerais
Other Study IDs: CAAE: 56548816.6.0000.5149
Record Dates: First submitted 2017-11-03; First posted 2017-11-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Nutritional Therapy Quality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nutritional status depletion is associated with complications such as increased morbidity and mortality, worsening of patients' quality of life and increased length of hospital stay. Thus, nutritional therapy defined as the set of therapeutic procedures for maintenance or recovery of the nutritional status of the patient, becomes a procedure of extreme importance in the hospital setting. It should be carried out by an interprofessional team, in order to ensure adequate patient care. Aim: This study intends to evaluate the reality of Nutritional Therapy in Brazil, 18 and 14 years after the introduction of the resolution n ° 272 and the RDC n ° 63, respectively, regarding the practice of this important therapy and the existence of interdisciplinary teams. Method: Descriptive, observational and national study. In each Brazilian state was selected the capital, and drawn a city of average and other one of small size. Next, a public, private and university hospital in each municipality was randomly selected. Data collection will be done by means of a questionnaire, based on the Secretary of Sanitary Surveillance of the Ministry of Health resolution n ° 272 and the RDC n ° 63. The questionnaire will be applied by the researchers, and directed to the health professionals involved in the Nutritional Therapy practice in each of the selected hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Hospitals with nutritional therapy

Exclusion Criteria:

* Hospitals with no nutritional therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitals with nutritional therapy (Public, private and teaching hospitals)
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The Reality of Nutritional Therapy in Brazil | December, 2017.
  The adequacy will be assessed using proper questionnaire prepared up from Resolution of Collegiate Board of the National Health Surveillance Agency Nº 63/2000 and portaria n° 272 of the Ministry of Health.

SECONDARY OUTCOMES:
Performance of interdisciplinary teams of nutritional therapy | December, 2017.
  The performance will be assessed using proper questionnaire prepared up from Resolution of Collegiate Board of the National Health Surveillance Agency Nº 63/2000 and portaria n° 272 of the Ministry of Health.
Number of patients in nutritional therapy in hospitals | December, 2017.
  Own Checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Clinics of the University Federal of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil